CLINICAL TRIAL: NCT04398602
Title: Leader and Team Performance During PPH Simulated Scenario: a Comparison Between Self- and Expert's Assessment
Brief Title: Leader and Team Performance During PPH Simulated Scenario
Status: Completed | Type: Observational
Sponsor: Capogna Giorgio (Other)
Responsible Party: Sponsor-Investigator, Capogna Giorgio, Director, EESOA Simulation Center, European e-Learning School in Obstetric Anesthesia
Organization: European e-Learning School in Obstetric Anesthesia (Other)
Other Study IDs: EESOA8
Record Dates: First submitted 2020-05-18; First posted 2020-05-21 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Obstetric Anesthesia Problems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: behavior of the leader — A study investigator, expert in both PPH and simulation debriefing, not involved in the simulation, observed each scenario to record and check the team's technical skills according to the established 23 PPH key tasks. The behavioral scores were assigned by two independent observers, experts in communication and evaluation in simulation, who reviewed the videos of each simulation each simulation all participants were asked to complete a survey related to the leader and the team behaviors. Questions required a yes/no answer or an answer based on an ordinal scale (1=poor, 5=excellent).
  Other Names: non technical skills performed by the team

SUMMARY:
The primary aim of this study is the progress of the performance of the leader and of the team for the postpartum hemorrhage (PPH) before and after four high-fidelity standardized scenarios of severe PPH (1500 mL blood loss) due to refractory uterine atony with anesthesia trainees.

DETAILED DESCRIPTION:
8 teams were studied: each team consisted of six participants, all anesthesia trainees, who were given the following roles for the scenario: senior anesthesiologist, anesthesia trainee, obstetrician, midwife, and nurse. The teams encountered the same scenario of a patient with atonic PPH following vaginal delivery. The scenario was repeated four times and the assigned roles to the participants, except that one of the senior anesthesiologists, rotated every each scenario.For the design of the PPH checklist, the authors reviewed PPH guidelines from recognized obstetric bodies (American College of Obstetricians and Gynecologists (ACOG) and the Royal College of Obstetricians and Gynaecologists), relevant papers from the literature and the investigator's institutional PPH protocol. The final action items for the checklist were selected by consensus by all authors. A standardized, 23 key tasks were identified for inclusion on the PPH checklist (non-behavioral skills) and this checklist worked as the reference guide for pre and post-workshop evaluation of the trainees.

For the design of the non-technical skills evaluation scores, the authors reviewed the non-technical skills evaluation instruments, such as the Anaesthetists' Non-Technical Skills (ANTS) behavioural marker system and the Ottawa Global Rating Scale (GRS). The final action items for the checklist were selected by consensus by all authors. Standardized, evaluation and self-evaluation questionnaires were developed .

No educational training was performed before the performance of the first scenario and participants were naïve to the scenario before performing each simulation.

All the teams underwent standardized educational training immediately before the second, third, and fourth scenarios. Every standardized educational training consisted of a 30 minutes session. At the beginning of the session, each participant was invited to write, in three minutes, on a piece of paper, what they would do in case of postpartum bleeding. Afterward each participant was invited to share and to write on the blackboard, one by one, on turn, the clinical procedures that he had previously reported in his personal paper. After this session the instructor, after having asked to all the participant whether there were something else to add, integrated, if necessary, the missing elements by using the 23 key tasks and reconfirmed the agreement with the group itself in order to have a shared check-list of the postpartum hemorrhage treatment.

The scenario consisted of a severe PPH (1500 mL blood loss) due to refractory uterine atony in a multiparous 28-year-old patient who had undergone a spontaneous vaginal delivery. The patient became tachycardic and hypotensive consistent with hemorrhagic shock. All simulations were performed in the simulation room using a high-fidelity mannequin (SinMom Maternal and Neonatal Birthing Simulator, Laerdal, Norway). All simulations were videotaped. The simulation was stopped when each team completed all 23 tasks of the checklist, or when 15 min had elapsed.

A study investigator, expert in both PPH and simulation debriefing, not involved in the simulation, observed each scenario to record and check the team's technical skills according to the established 23 PPH key tasks. The behavioral scores were assigned by two independent observers, experts in communication and evaluation in simulation, who reviewed the videos of each simulation. After each simulation all participants were asked to complete a survey related to the leader and the team behaviors. Questions required a yes/no answer or an answer based on an ordinal scale (1=poor, 5=excellent). Survey questions are presented in the Appendix

ELIGIBILITY:
Inclusion Criteria:

* anesthesia trainee

Exclusion Criteria:

* none

Ages: 25 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: anesthesia trainees
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
leader behavior | 15 minutes
  The behavioral scores (Likert Scale)) were assigned by two independent observers, experts in communication and evaluation in simulation, who reviewed the videos of each simulation.
team performance | 15 minutes
  A study investigator, expert in both PPH and simulation debriefing, not involved in the simulation, observed each scenario to record and check the team's technical skills according to the established 23 PPH key task.
leader self assessment | 15 minutes
  After each simulation all the leaders were asked to complete a survey related to the leader and the team behaviors. Questions required a yes/no answer or an answer based on an ordinal scale (1=poor, 5=excellent).
team self assessment | 15 minutes
  After each simulation all participants were asked to complete a survey related to the leader and the team behaviors. Questions required a yes/no answer or an answer based on an ordinal scale (1=poor, 5=excellent).

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Capogna, MD, Study Director — European e-Learning School in Obstetric Anesthesia
Locations (1):
- Eesoa Simulation Center, Roma, Italy

IPD SHARING:
Plan to Share IPD: No